CLINICAL TRIAL: NCT03009578
Title: Intravenous Iron Sucrose Versus Oral Ferrous Bis-glycinate for Treatment of Postpartum Iron Deficiency Anemia: a Randomized Clinical Trial
Brief Title: Iron Sucrose Versus Ferrous Bis-glycinate for Treatment of Iron Deficiency Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OFB-IDA
Record Dates: First submitted 2017-01-02; First posted 2017-01-04 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Ferric Oxide, Saccharated; ferrous bisglycinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous iron (Experimental): Women will receive iron sucrose (sacrofer ampules 100 mg/5ml) A patient's total body iron deficit will be calculated using the Ganzoni formula (total iron dose = [body weight (kilogram)× (15-actual Hemoglobin)] × 2.4 + 500 mg) then the total dose will be divided on 3 settings
  Interventions: Drug: Iron Sucrose Injection
- Oral ferrous bis-glycinate (Active Comparator): Women will receive oral ferrous bis-glycinate fully reacted amino acid 27 mg tablets
  Interventions: Drug: Ferrous Bisglycinate

INTERVENTIONS:
Drug: Iron Sucrose Injection — iron Intramuscular injections
  Arms: Intravenous iron
Drug: Ferrous Bisglycinate — oral iron tablets
  Arms: Oral ferrous bis-glycinate

SUMMARY:
Iron deficiency may result from inadequate dietary intake, achlorhydria or excessive ingestion of proton pump inhibitors, parasitic infestations, chronic infections and repeated pregnancies. Iron supplementation of antenatal patients is a basic tenet of antenatal care programmes in numerous developing and underdeveloped nations.

Postpartum anemia is defined as hemoglobin of less than 11.5 gm% during the postpartum period. The prevalence of postpartum anemia varies from 4 - 27%. Chronic iron deficiency due to inadequate intake/ lack of iron supplementation during pregnancy, repeated pregnancies and postpartum hemorrhage are important causes of postpartum anemia

ELIGIBILITY:
Inclusion Criteria:

Hemoglobin level 7-11.5 gm/dl. No chronic diseases. Breastfeeding. Delivered at gestational age >38 weeks. Within 24-72 hours postpartum. Women who accept to participate in the study

Exclusion Criteria:

1. Severe anemia < 7 gm/dl.
2. Women received iron therapy during pregnancy.
3. Intolerance to iron preparations
4. Anemia due to other causes
5. Peripartum blood transfusion.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
the percentage of patients achieving Hb rise 3 gm or more | 6 weeks

SECONDARY OUTCOMES:
Mean rise of Hb from baseline to 6 weeks. | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided